CLINICAL TRIAL: NCT02976688
Title: Effects of Short-chain Fatty Acids, Here Sodium Propionate, a Metabolism Product of the Human Gut-microbiome, on Inflammatory and Metabolic Parameters in Patients on Maintenance Hemodialysis - a Pilot Study
Brief Title: Effects of Short-chain Fatty Acids on Inflammatory and Metabolic Parameters in Maintenance Hemodialysis
Acronym: PLAN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria ASL Avellino 2 (Other)
Responsible Party: Principal Investigator, Dr Biagio Di Iorio, Dr, Chief Nephrology Division, Azienda Sanitaria ASL Avellino 2
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASL AVELLINO
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Endstage Renal Disease
Keywords: Endstage renal Disease; Hemodialysis
MeSH Terms: interventions — sodium propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium propionate (Experimental): Sodium propionate will be administered with a daily intake of 2 x 500 mg in form of capsules for 12 weeks.
  Interventions: Other: Sodium Propionate

INTERVENTIONS:
Other: Sodium Propionate — Sodium propionate is a non-toxic food additive, confirmed and licensed by the European Food Safety Authority (EFSA) sodium propionate E281. We are planning the oral application of 500 mg SP 2x per day. This dose is about 0.014 mg/kg of the body weight. Therefore, no risk of toxicity is expected in the patients.
  Other Names: Sodium propionate E281

SUMMARY:
End-stage renal disease (ESRD) is associated with multiple comorbidities such as cardiovascular disease, anemia, mineral and bone disorders, malnutrition, body wasting, muscle loss (sarcopenia), neurological problems and infections resulting in a poor survival.

In the pathogenesis of the uremic syndrome the altered intestinal function seems to be an important contributor. While the normal gut microbiota plays a prominent role in the maintenance of health and disease prevention, changes of its composition is associated with numerous diseases such as obesity, type 2 diabetes, cardiovascular disturbances and auto-immune diseases.In ESRD metabolic alterations of uremia results in quantitative and qualitative changes of its bacterial flora with an overgrowth of pathobionts (1). Due to concomitant disruption of the intestinal barrier function, noxious luminal products are translocated in the body's internal milieu (2).The accumulation of these compounds correlates with systemic inflammation, protein wasting and accelerated cardiovascular complications in hemodialysis patients (3).

Short-chain fatty acids (SCFA) are produced in the colon and distal small intestine by anaerobic bacteria following fermentation of complex carbohydrates.They have been shown to exert anti-inflammatory, anti-cancer, antibacterial and antidiabetic effects (4). Supplementation of SCFA exerts anti-inflammatory actions both in intestinal epithelial cells (5) and in the cardiovascular system (6). They also positively influence auto- immune reactions /diseases (7,8).

In this study we want to investigate in MHD patients whether a treatment with SCFA in form of sodium propionate (SP) modulates the systemic inflammation, insulin resistance and accumulation of intestinal uremic toxins.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is associated with multiple comorbidities such as cardiovascular disease, anemia, mineral and bone disorders, malnutrition, body wasting, muscle loss (sarcopenia), neurological problems and infections resulting in a poor survival. Important promoters of these obstacles are enhanced generation of reactive oxygen species (ROS), systemic inflammation, acquired immunodeficiency (9, 10) and an impaired glucose and insulin homeostasis (11).

Systemic inflammation and oxidative stress in ESRD are induced by activation of the innate immune system involving monocytes, macrophages, granulocytes and cellular constituents (endothelial cell activation) as well as depletion of natural regulatory T cells that impairs their ability to suppress inflammation .The concomitant reduced humoral immunity is favored by depletion of antigen presenting dendritic cells, a lowered CD44/CD8 T cell ratio, depletion of naïve and central memory T cells, diffuse B cell lymphopenia and an impaired phagocytic ability of monocytes and PMNs (12).

Insulin resistance (IR) participates in the pathogenesis of multiple metabolic and cardiovascular disturbances (13) and is an important factor of the accelerated muscle protein degradation in ESRD (14). Underlying mechanisms of IR are the metabolic inflammation, in particular elevated LPS levels.

In the pathogenesis of the uremic syndrome the altered intestinal function seems to be an important contributor. While the normal gut microbiota plays a prominent role in the maintenance of health and disease prevention, changes of its composition is associated with numerous diseases such as obesity, type 2 diabetes, cardiovascular disturbances and auto-immune diseases. In ESRD metabolic alterations of uremia results in quantitative and qualitative changes of its bacterial flora with an overgrowth of pathobionts (1). Due to concomitant disruption of the intestinal barrier function, noxious luminal products are translocated in the body's internal milieu (Fig.2). The passage includes whole bacteria (going into mesenteric lymph nodes), endotoxins/ lipoproteinlipase (LPS) (cell wall components of the bacteria) and other noxious luminal products which induce a persistent local (gut) and systemic inflammation.The process is intensified by the intestinal generation of several pro-inflammatory uremic toxins such as indoxyl sulfate, p-cresyl sulfate and trimethyamine-N-oxide (2).The accumulation of these compounds correlates with systemic inflammation, protein wasting and accelerated cardiovascular complications in hemodialysis patients (3).

Short-chain fatty acids (SCFA) are produced in the colon and distal small intestine by anaerobic bacteria following fermentation of complex carbohydrates. The 3 major compounds are acetic acid, butyric and propionic acids. SCFA contribute to the health of the gut (microbiome and mucosa) and the host. They have been shown to exert anti-inflammatory, anti-cancer, antibacterial and antidiabetic effects. Lower values and an dysbiotic gut contribute to various diseases such colitis, type 2 diabetes, rheumatoid disease and multiple sclerosis. Supplementation of SCFA exerts anti-inflammatory actions both in intestinal epithelial cells (5) and in the cardiovascular system (6). They also positively influence auto- immune reactions /diseases (7, 8). In particular SCFA enhances formation of regulatory T cells in the colon which are critical for regulating intestinal inflammation (15). Also effector T cells such as Il-10 are implicated (16). Likewise SCFA are involved in the control of body weight and insulin sensitivity (17), cholesterol synthesis (18) and retardation of progressive CKD.

In patients on maintenance hemodialysis (MHD) a diet with a high fiber content, which favors the intestinal SCFA formation (19), lowered the plasma levels of the colon-derived solutes indoxyl sulfate and possibly p-cresol sulfate (20) and reduced inflammation, cardiovascular diseases and all-cause mortality in CKD/ESRD patients (21). However, in ESRD consumption of a fiber rich diet is limited due to the risk of hyperpotassemia. In addition the frequent antibiotic therapy, application of phosphate binder or iron therapy alters the gut microbiome.

The following mechanisms have been proposed for the actions of SCFA: the G-protein-coupled receptors GPR 41 and GPR 43 (the free fatty acid receptors FFAR 3 and 2 ), GPR 109a, Olfr78 , the inhibition of histone deacetylases (HDAC) and stimulation of histone acetyltransferase (HAT) activity (22, 23).

n this study we want to investigate in MHD patients whether a treatment with SCFA in form of sodium propionate (SP) modulates the systemic inflammation, insulin resistance and accumulation of intestinal uremic toxins. SP is chemically composed by a carboxylic acid moiety and a small hydrocarbon chain with three carbon atoms (black balls), two oxygen (red balls) and the white hydrogen atoms.

SP is involved in most effects of the short chain fatty acids including inhibition of intestinal and hepatocyte lipid synthesis (24), lowering of fasting glycemia (25, 26) and protection against diet-induced obesity ( 27). SP also regulates colonic T-reg cell homeostasis (28) and exerts marked anti-inflammatory actions including intestinal epithelial cells and macrophages (29) as well as in neutrophils, colon cells and colon cultures (30). It improved experimental autoimmune encephalomyelitis (31) and experimental acute renal failure (32). In addition antibacterial effects were documented (33, 34).

The patients under maintenance hemodialysis will receive the food additive sodium propionate with a daily intake of 2 x 500 mg in form of capsules (Propicum) for 12 weeks. The demographic information and the blood chemistry will be collected before the study, after 6, 12 and 16 weeks of drug administration.

The project will last for one year. The planned patient group should comprise of 15 patients on maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Stable hemodialysis patients treated by renal replacement therapy for at least 6 months
* Written informed consent written

Exclusion Criteria:

* Patients with malnutrition, infections, carcinoma, previous renal transplant, intestinal diseases (medically diagnosed irritable bowel syndrome, Crohn's disease, ulcerative colitis and diarrhea) and antibiotic treatment within one month of study will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Variation from the beginning to the study end of serum inflammatory biomarkers | 16 weeks
  endotoxin /lipopolysaccharide levels, high sensitivity C-reactive protein (hs-CRP), fibrinogen, interleukin 6 (IL-6), tumor necrosis factor α (TNF-α), IL-10, IL-2, INFγ, TGFβ, IL-4, IL-1β, IL-17a and white blood cell count.
Variation from the beginning to the study end of serum oxidative stress biomarkers | 16 weeks
  glutathione peroxidase, malone dialdehyde
Variation from the beginning to the study end of insulin resistance | 16 weeks
  Determination of Homa Index (Homeostasis Model Assessment) by measurement fasting blood sugar and insulin level as well as hemoglobin HbA1c. IR appears to be as associated of metabolic disorders including lipid abnormalities, atherosclerotic cardiovascular disease and accelerated muscle protein degradation (Wang et al. 2006). IL is induced in particular by systemic inflammation.
Variation from the beginning to the study end of serum lipid levels | 16 weeks
  Triglycerides, total cholesterol, high and low density cholesterol
Variation from the beginning to the study end of hormonal parameter | 16 weeks
  Leptin, resistin, adiponectin and glucagon-like peptide -1.
Variation from the beginning to the study end of uremic toxins produced in the intestinal tract | 16 weeks
  p-cresyl sulfate, indoxyl sulfate and trimethylamine -N-oxide
Variation from the beginning to the study end of nutritional status | 16 weeks
  Serum albumin
Variation from the beginning to the study end of parameters of well-being | 16 weeks
  patient reported health (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Di Iorio, Chief, PhD, Principal Investigator — ASL AVELLINO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469
- [Background] Aronov PA, Luo FJ, Plummer NS, Quan Z, Holmes S, Hostetter TH, Meyer TW. Colonic contribution to uremic solutes. J Am Soc Nephrol. 2011 Sep;22(9):1769-76. doi: 10.1681/ASN.2010121220. Epub 2011 Jul 22. PMID 21784895
- [Background] Barreto FC, Barreto DV, Liabeuf S, Meert N, Glorieux G, Temmar M, Choukroun G, Vanholder R, Massy ZA; European Uremic Toxin Work Group (EUTox). Serum indoxyl sulfate is associated with vascular disease and mortality in chronic kidney disease patients. Clin J Am Soc Nephrol. 2009 Oct;4(10):1551-8. doi: 10.2215/CJN.03980609. Epub 2009 Aug 20. PMID 19696217
- [Background] Ramezani A, Raj DS. The gut microbiome, kidney disease, and targeted interventions. J Am Soc Nephrol. 2014 Apr;25(4):657-70. doi: 10.1681/ASN.2013080905. Epub 2013 Nov 14. PMID 24231662
- [Background] Iraporda C, Errea A, Romanin DE, Cayet D, Pereyra E, Pignataro O, Sirard JC, Garrote GL, Abraham AG, Rumbo M. Lactate and short chain fatty acids produced by microbial fermentation downregulate proinflammatory responses in intestinal epithelial cells and myeloid cells. Immunobiology. 2015 Oct;220(10):1161-9. doi: 10.1016/j.imbio.2015.06.004. Epub 2015 Jun 10. PMID 26101138
- [Background] Vinolo MA, Rodrigues HG, Nachbar RT, Curi R. Regulation of inflammation by short chain fatty acids. Nutrients. 2011 Oct;3(10):858-76. doi: 10.3390/nu3100858. Epub 2011 Oct 14. PMID 22254083
- [Background] Maslowski KM, Vieira AT, Ng A, Kranich J, Sierro F, Yu D, Schilter HC, Rolph MS, Mackay F, Artis D, Xavier RJ, Teixeira MM, Mackay CR. Regulation of inflammatory responses by gut microbiota and chemoattractant receptor GPR43. Nature. 2009 Oct 29;461(7268):1282-6. doi: 10.1038/nature08530. PMID 19865172
- [Background] Richards JL, Yap YA, McLeod KH, Mackay CR, Marino E. Dietary metabolites and the gut microbiota: an alternative approach to control inflammatory and autoimmune diseases. Clin Transl Immunology. 2016 May 13;5(5):e82. doi: 10.1038/cti.2016.29. eCollection 2016 May. PMID 27350881
- [Background] Vaziri ND. Oxidative stress in uremia: nature, mechanisms, and potential consequences. Semin Nephrol. 2004 Sep;24(5):469-73. doi: 10.1016/j.semnephrol.2004.06.026. PMID 15490413
- [Background] Anders HJ, Andersen K, Stecher B. The intestinal microbiota, a leaky gut, and abnormal immunity in kidney disease. Kidney Int. 2013 Jun;83(6):1010-6. doi: 10.1038/ki.2012.440. Epub 2013 Jan 16. PMID 23325079
- [Background] de Boer IH, Zelnick L, Afkarian M, Ayers E, Curtin L, Himmelfarb J, Ikizler TA, Kahn SE, Kestenbaum B, Utzschneider K. Impaired Glucose and Insulin Homeostasis in Moderate-Severe CKD. J Am Soc Nephrol. 2016 Sep;27(9):2861-71. doi: 10.1681/ASN.2015070756. Epub 2016 Jan 28. PMID 26823551
- [Background] Vaziri ND, Pahl MV, Crum A, Norris K. Effect of uremia on structure and function of immune system. J Ren Nutr. 2012 Jan;22(1):149-56. doi: 10.1053/j.jrn.2011.10.020. PMID 22200433
- [Background] DeFronzo RA, Ferrannini E. Insulin resistance. A multifaceted syndrome responsible for NIDDM, obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Diabetes Care. 1991 Mar;14(3):173-94. doi: 10.2337/diacare.14.3.173. PMID 2044434
- [Background] Wang X, Hu Z, Hu J, Du J, Mitch WE. Insulin resistance accelerates muscle protein degradation: Activation of the ubiquitin-proteasome pathway by defects in muscle cell signaling. Endocrinology. 2006 Sep;147(9):4160-8. doi: 10.1210/en.2006-0251. Epub 2006 Jun 15. PMID 16777975
- [Background] Smith PM, Howitt MR, Panikov N, Michaud M, Gallini CA, Bohlooly-Y M, Glickman JN, Garrett WS. The microbial metabolites, short-chain fatty acids, regulate colonic Treg cell homeostasis. Science. 2013 Aug 2;341(6145):569-73. doi: 10.1126/science.1241165. Epub 2013 Jul 4. PMID 23828891
- [Background] Park J, Kim M, Kang SG, Jannasch AH, Cooper B, Patterson J, Kim CH. Short-chain fatty acids induce both effector and regulatory T cells by suppression of histone deacetylases and regulation of the mTOR-S6K pathway. Mucosal Immunol. 2015 Jan;8(1):80-93. doi: 10.1038/mi.2014.44. Epub 2014 Jun 11. PMID 24917457
- [Background] Canfora EE, Jocken JW, Blaak EE. Short-chain fatty acids in control of body weight and insulin sensitivity. Nat Rev Endocrinol. 2015 Oct;11(10):577-91. doi: 10.1038/nrendo.2015.128. Epub 2015 Aug 11. PMID 26260141
- [Background] Hara H, Haga S, Aoyama Y, Kiriyama S. Short-chain fatty acids suppress cholesterol synthesis in rat liver and intestine. J Nutr. 1999 May;129(5):942-8. doi: 10.1093/jn/129.5.942. PMID 10222383
- [Background] Psichas A, Sleeth ML, Murphy KG, Brooks L, Bewick GA, Hanyaloglu AC, Ghatei MA, Bloom SR, Frost G. The short chain fatty acid propionate stimulates GLP-1 and PYY secretion via free fatty acid receptor 2 in rodents. Int J Obes (Lond). 2015 Mar;39(3):424-9. doi: 10.1038/ijo.2014.153. Epub 2014 Aug 11. PMID 25109781
- [Background] Sirich TL, Plummer NS, Gardner CD, Hostetter TH, Meyer TW. Effect of increasing dietary fiber on plasma levels of colon-derived solutes in hemodialysis patients. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1603-10. doi: 10.2215/CJN.00490114. Epub 2014 Aug 21. PMID 25147155
- [Background] Krishnamurthy VM, Wei G, Baird BC, Murtaugh M, Chonchol MB, Raphael KL, Greene T, Beddhu S. High dietary fiber intake is associated with decreased inflammation and all-cause mortality in patients with chronic kidney disease. Kidney Int. 2012 Feb;81(3):300-6. doi: 10.1038/ki.2011.355. Epub 2011 Oct 19. PMID 22012132
- [Background] Brown AJ, Goldsworthy SM, Barnes AA, Eilert MM, Tcheang L, Daniels D, Muir AI, Wigglesworth MJ, Kinghorn I, Fraser NJ, Pike NB, Strum JC, Steplewski KM, Murdock PR, Holder JC, Marshall FH, Szekeres PG, Wilson S, Ignar DM, Foord SM, Wise A, Dowell SJ. The Orphan G protein-coupled receptors GPR41 and GPR43 are activated by propionate and other short chain carboxylic acids. J Biol Chem. 2003 Mar 28;278(13):11312-9. doi: 10.1074/jbc.M211609200. Epub 2002 Dec 19. PMID 12496283
- [Background] Correa-Oliveira R, Fachi JL, Vieira A, Sato FT, Vinolo MA. Regulation of immune cell function by short-chain fatty acids. Clin Transl Immunology. 2016 Apr 22;5(4):e73. doi: 10.1038/cti.2016.17. eCollection 2016 Apr. PMID 27195116
- [Background] Wright RS, Anderson JW, Bridges SR. Propionate inhibits hepatocyte lipid synthesis. Proc Soc Exp Biol Med. 1990 Oct;195(1):26-9. doi: 10.3181/00379727-195-43113. PMID 2399259
- [Background] Boillot J, Alamowitch C, Berger AM, Luo J, Bruzzo F, Bornet FR, Slama G. Effects of dietary propionate on hepatic glucose production, whole-body glucose utilization, carbohydrate and lipid metabolism in normal rats. Br J Nutr. 1995 Feb;73(2):241-51. doi: 10.1079/bjn19950026. PMID 7718543
- [Background] Puddu A, Sanguineti R, Montecucco F, Viviani GL. Evidence for the gut microbiota short-chain fatty acids as key pathophysiological molecules improving diabetes. Mediators Inflamm. 2014;2014:162021. doi: 10.1155/2014/162021. Epub 2014 Aug 17. PMID 25214711
- [Background] Arora T, Loo RL, Anastasovska J, Gibson GR, Tuohy KM, Sharma RK, Swann JR, Deaville ER, Sleeth ML, Thomas EL, Holmes E, Bell JD, Frost G. Differential effects of two fermentable carbohydrates on central appetite regulation and body composition. PLoS One. 2012;7(8):e43263. doi: 10.1371/journal.pone.0043263. Epub 2012 Aug 29. PMID 22952656
- [Background] Zeng X, Sunkara LT, Jiang W, Bible M, Carter S, Ma X, Qiao S, Zhang G. Induction of porcine host defense peptide gene expression by short-chain fatty acids and their analogs. PLoS One. 2013 Aug 30;8(8):e72922. doi: 10.1371/journal.pone.0072922. eCollection 2013. PMID 24023657
- [Background] Tedelind S, Westberg F, Kjerrulf M, Vidal A. Anti-inflammatory properties of the short-chain fatty acids acetate and propionate: a study with relevance to inflammatory bowel disease. World J Gastroenterol. 2007 May 28;13(20):2826-32. doi: 10.3748/wjg.v13.i20.2826. PMID 17569118
- [Background] Haghikia A, Jorg S, Duscha A, Berg J, Manzel A, Waschbisch A, Hammer A, Lee DH, May C, Wilck N, Balogh A, Ostermann AI, Schebb NH, Akkad DA, Grohme DA, Kleinewietfeld M, Kempa S, Thone J, Demir S, Muller DN, Gold R, Linker RA. Dietary Fatty Acids Directly Impact Central Nervous System Autoimmunity via the Small Intestine. Immunity. 2015 Oct 20;43(4):817-29. doi: 10.1016/j.immuni.2015.09.007. PMID 26488817
- [Background] Andrade-Oliveira V, Amano MT, Correa-Costa M, Castoldi A, Felizardo RJ, de Almeida DC, Bassi EJ, Moraes-Vieira PM, Hiyane MI, Rodas AC, Peron JP, Aguiar CF, Reis MA, Ribeiro WR, Valduga CJ, Curi R, Vinolo MA, Ferreira CM, Camara NO. Gut Bacteria Products Prevent AKI Induced by Ischemia-Reperfusion. J Am Soc Nephrol. 2015 Aug;26(8):1877-88. doi: 10.1681/ASN.2014030288. Epub 2015 Jan 14. PMID 25589612
- [Background] Hung CC, Garner CD, Slauch JM, Dwyer ZW, Lawhon SD, Frye JG, McClelland M, Ahmer BM, Altier C. The intestinal fatty acid propionate inhibits Salmonella invasion through the post-translational control of HilD. Mol Microbiol. 2013 Mar;87(5):1045-60. doi: 10.1111/mmi.12149. Epub 2013 Jan 28. PMID 23289537
- [Background] Sunkara LT, Jiang W, Zhang G. Modulation of antimicrobial host defense peptide gene expression by free fatty acids. PLoS One. 2012;7(11):e49558. doi: 10.1371/journal.pone.0049558. Epub 2012 Nov 15. PMID 23166711